CLINICAL TRIAL: NCT00077467
Title: A Phase I Study of PS-341 (Velcade, Bortezomib) in Pediatric Patients With Refractory/Recurrent Leukemias
Brief Title: Bortezomib in Treating Young Patients With Refractory or Recurrent Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01809; ADVL0317; CDR0000350340; COG-ADVL0317; U01CA097452 (NIH)
Record Dates: First submitted 2004-02-10; First posted 2004-02-12 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Blastic Phase Chronic Myelogenous Leukemia; Childhood Acute Promyelocytic Leukemia (M3); Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia
MeSH Terms: conditions — Blast Crisis; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Bortezomib

ARMS (1):
- Arm I (Experimental): Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: bortezomib; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of bortezomib in treating young patients with refractory or recurrent leukemia. Bortezomib may stop the growth of cancer cells by blocking the enzymes necessary for their growth.

DETAILED DESCRIPTION:
OBJECTIVES: Primary I. Determine the maximum tolerated dose and recommended phase II dose of bortezomib in children with refractory or recurrent leukemia.

II. Determine the toxic effects of this drug in these patients. III. Determine the pharmacokinetics of this drug in these patients.

Secondary I. Determine, preliminarily, the antitumor activity of this drug in these patients.

II. Determine, preliminarily, the biologic activity of this drug in these patients.

OUTLINE: This is a dose-escalation, open-label, multicenter study.

Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of bortezomib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A total of 3-36 patients will be accrued for this study within 1.5-36 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed leukemia of 1 of the following types:

  * Acute lymphoblastic leukemia
  * Acute myeloid leukemia
  * Chronic myelogenous leukemia in blast crisis
* Relapsed or refractory disease
* Immunophenotypically confirmed disease, either at initial diagnosis or relapse
* More than 25% blasts in the bone marrow (M3 bone marrow)
* Active extramedullary disease (except leptomeningeal disease) allowed
* No known curative therapy or therapy proven to prolong survival with an acceptable quality of life available
* Performance status - Karnofsky 50-100% (for patients age 11 to 21)
* Performance status - Lansky 50-100% (for patients age 10 and under)
* Platelet count ≥ 20,000/mm^3*
* Hemoglobin ≥ 8.0 g/dL*
* WBC < 20,000/mm^3** (hydroxyurea for cytoreduction allowed)
* No hyperleukocytosis (i.e., WBC > 100,000/mm^3)
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT ≤ 5 times ULN
* Albumin ≥ 2 g/dL
* Creatinine clearance or radioisotope glomerular filtration rate ≥ 70 mL/min
* Creatinine based on age as follows:

  * ≤ 0.8 mg/dL for patients age 5 and under
  * ≤ 1.0 mg/dL for patients age 6 to 10
  * ≤ 1.2 mg/dL for patients age 11 to 15
  * ≤ 1.5 mg/dL for patients age 16 to 21
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled infection
* Recovered from prior immunotherapy
* At least 7 days since prior filgrastim (G-CSF) or sargramostim (GM-CSF)
* At least 7 days since prior biologic agents
* At least 3 months since prior stem cell transplantation or rescue and no evidence of active graft-versus-host disease
* No concurrent prophylactic G-CSF during course 1 of study
* No concurrent immunotherapy
* No concurrent biologic therapy
* Recovered from prior chemotherapy
* At least 24 hours since prior hydroxyurea for cytoreduction
* At least 6 weeks since prior nitrosoureas
* No concurrent chemotherapy
* At least 7 days since prior steroids (except as premedication prior to blood product transfusion)
* Recovered from prior radiotherapy
* At least 2 weeks since prior small port local palliative radiotherapy
* At least 3 months since prior total body irradiation, craniospinal irradiation, or irradiation to more than 50% of the pelvis
* At least 6 weeks since other prior substantial bone marrow radiotherapy
* No concurrent radiotherapy
* At least 7 days since prior retinoids
* No other concurrent investigational agents
* No other concurrent anticancer agents
* No concurrent anticonvulsant medications known to activate the cytochrome p450 system (e.g., phenytoin, carbamazepine, or phenobarbital)

  * Concurrent benzodiazepines and gabapentin are allowed

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2004-01; Primary Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose and recommended phase II dose | Up to 21 days
Toxicity as assessed by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) 3.0 | Up to 2 years
Pharmacokinetics as assessed by confidence intervals (CI), area under the curve (AUC), and half-life (T ½) | Pretreatment, days 1, 8, 18-22 of course 1

SECONDARY OUTCOMES:
Antitumor activity | Up to 2 years
Correlate apoptosis and NF-kB activation | Prestudy, days 8 and 18

CONTACTS AND LOCATIONS:
Overall Officials: Terzah Horton, Principal Investigator — COG Phase I Consortium
Locations (1):
- COG Phase I Consortium, Arcadia, California, United States